CLINICAL TRIAL: NCT06497504
Title: A Multicenter, Randomized, Double-Blind, Placebo-controlled Study to Assess the Efficacy and Safety of Treatment With Bepirovirsen in Participants Living With Human Immunodeficiency Virus and Chronic Hepatitis B Virus Infection on Antiretroviral Treatment
Brief Title: Study of Bepirovirsen in Participants Living With Human Immunodeficiency Virus and Chronic Hepatitis B Virus Infection (B-Focus)
Acronym: B-Focus
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 219231; 2023-509588-25 (Other: EU CT Number)
Record Dates: First submitted 2024-07-05; First posted 2024-07-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hepatitis B
Keywords: Antiretroviral treatment; Bepirovirsen; Human immunodeficiency virus; Hepatitis B virus; Placebo
MeSH Terms: conditions — Hepatitis B; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants receiving Bepirovirsen (Experimental): Participants will receive bepirovirsen.
  Interventions: Drug: Bepirovirsen
- Participants receiving Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bepirovirsen — Bepirovirsen will be administered.
  Arms: Participants receiving Bepirovirsen
Drug: Placebo — Placebo will be administered.
  Arms: Participants receiving Placebo

SUMMARY:
This study will evaluate the efficacy and safety of bepirovirsen compared to placebo in participants with human immunodeficiency virus (HIV)/hepatitis B virus (HBV) co-infection.

ELIGIBILITY:
Inclusion Criteria:

1. Documented chronic hepatitis B virus (HBV) infection and documented human immunodeficiency virus (HIV)-1 infection greater than equal to (>=) 12 months prior to Screening.
2. Must be on uninterrupted antiretroviral therapy (ART) containing at least tenofovir disoproxil (TDF) or tenofovir alafenamide (TAF) plus lamivudine (3TC) or emtricitabine (FTC) for greater than (>)12 months, with no planned changes to the stable regimen over the duration of the study.

   o Switch in ART is permitted >=6 months prior to Screening for reasons not related to loss of HIV or HBV control (e.g., change in formulary, tolerability, side effects).
3. Documented evidence of at least 2 plasma HIV-1 ribonucleic acid (RNA) measurements less than (<) 50 copies per milliliter (copies/mL) are required in the 12 months prior to Screening: 1 within 6 to 12 months prior to Screening and 1 within 6 months prior to Screening.
4. Plasma or serum HBV deoxyribonucleic acid (DNA) concentration must be adequately suppressed, defined as plasma or serum HBV DNA <90 international units per milliliter (IU/mL).
5. Plasma or serum HBsAg concentration >100 IU/mL and <=3000 IU/mL.
6. Plasma HIV-1 RNA concentration must be undetectable, defined as plasma HIV 1 RNA <50 copies/mL.
7. Cluster of differentiation 4 (CD4) count >=350 cells per cubic millimeter (cells/mm^3).
8. Alanine aminotransferase (ALT) <=2 times upper limit of normal (ULN).

Exclusion Criteria:

1. History of or suspected liver cirrhosis and/or evidence of cirrhosis.
2. Diagnosed or suspected hepatocellular carcinoma (HCC).
3. History of extrahepatic disorders possibly related to HBV immune conditions (e.g., nephrotic syndrome, any type of glomerulonephritis, polyarteritis nodosa, cryoglobulinemia, uncontrolled hypertension).
4. Coinfection with:

   1. Hepatitis C virus (HCV) with positive HCV antibody and detectable HCV RNA at Screening.

      I. HCV treatment should have completed >12 months prior to Screening.
   2. Hepatitis D virus (HDV) defined as positive or equivocal HDV antibody regardless of HDV RNA level.
5. Clinically significant abnormalities, aside from HIV-1 infection and chronic HBV infection in medical history (e.g., moderate severe liver disease other than chronic HBV/HIV, acute coronary syndrome within 6 months of Screening, major surgery within 3 months of Screening, significant/unstable cardiac disease, uncontrolled diabetes, bleeding diathesis coagulopathy) or clinically significant physical examination findings.
6. Untreated syphilis infection (positive rapid plasma reagin [RPR] at Screening without clear documentation of treatment) are excluded unless they complete treatment during the Screening period and 7 days prior to randomization.
7. History of malignancy within the past 5 years with the exception of specific cancers that are cured by surgical resection (e.g., skin cancer). Participants under evaluation for possible malignancy are not eligible.
8. History of vasculitis or presence of symptoms and signs of potential vasculitis (e.g., vasculitic rash, skin ulceration, repeated blood detected in urine without identified cause), current or history of an autoimmune condition or history/presence of other diseases that may be associated with vasculitis condition (e.g., systemic lupus erythematosus, rheumatoid arthritis, relapsing polychondritis, mononeuritis multiplex).
9. Participants who in the investigator's judgment, have a significant risk of suicide or self-harm.
10. Alcohol or drug abuse/dependence
11. Currently taking, or took within 3 months of Screening, any immunosuppressing drugs (e.g., prednisone), other than a short course of therapy (<=2 weeks) or topical/inhaled steroid use.
12. Participants to whom immunosuppressive treatment, including therapeutic doses of steroids, is contraindicated should not be considered for enrolment in the study.
13. Currently taking, or has taken within 12 months of Screening, any interferon containing therapy.
14. Participants requiring anti coagulation therapies (e.g., warfarin, Factor Xa inhibitors) or anti platelet agents (including but not limited to clopidogrel or aspirin) unless treatment can safely be discontinued throughout duration of study intervention, by the discretion of the investigator. Occasional use is permitted.
15. Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
16. Prior treatment with any oligonucleotide or small interfering ribonucleic acid (siRNA) within 12 months prior to the first dosing day.
17. Prior treatment with bepirovirsen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2027-04-22 (Estimated); Study Completion 2027-04-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving hepatitis B virus (HBV) virologic response at 36 weeks after scheduled end of study treatment in absence of rescue medication | At study week 60
  HBV virologic response defined as HBV surface antigen (HBsAg) not detected and HBV deoxyribonucleic acid (DNA) less than (<) lower limit of quantification (LLOQ).

SECONDARY OUTCOMES:
Percentage of participants achieving HBV virologic response at the scheduled end of study treatment in absence of rescue medication | At study week 24
  HBV virologic response defined as HBsAg not detected and HBV DNA <LLOQ.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (41):
- United States (7):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Hillsborough, New Jersey
- Argentina (4):
  - GSK Investigational Site, Almagro
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, Rosario
- Brazil (6):
  - GSK Investigational Site, Aracaju
  - GSK Investigational Site, Campinas
  - GSK Investigational Site, Curitiba
  - GSK Investigational Site, Manaus
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São Paulo
- Canada (4):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- France (5):
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Melun
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
- Italy (5):
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Sassari
- South Africa (3):
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Reiger Park
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Madrid
- Taiwan (2):
  - GSK Investigational Site, Banchiau Taipei
  - GSK Investigational Site, Kaohsiung City
- United Kingdom (2):
  - GSK Investigational Site, Bristol Avon
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/